CLINICAL TRIAL: NCT03426657
Title: First-line Treatment of Locally Advanced HNSCC With Double Checkpoint Blockade and Radiotherapy Dependent on Intratumoral CD8+ T Cell Infiltration (CheckRad-CD8, EudraCT NUMBER: 2017-003226-33)
Brief Title: Radiotherapy With Double Checkpoint Blockade of Locally Advanced HNSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CheckRad-CD8
Record Dates: First submitted 2018-01-24; First posted 2018-02-08 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Prospective, Open-Label, Non-Randomized
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Tremelimumab + RT (Experimental): Durvalumab (1500 mg,q4W) + Tremelimumab (75 mg, q4W / since Amendment 3: 300 mg absolute dose d5) for up to a maximum of 4 doses/cycles combined with radiotherapy (35 x 2.0/1.8/1.6 Gy) followed by durvalumab monotherapy 1500mg via IV infusion q4W, starting 4 weeks after the last infusion of the combination, for up to a maximum of 8 additional durvalumab doses.
  Interventions: Combination Product: Durvalumab + Tremelimumab + RT

INTERVENTIONS:
Combination Product: Durvalumab + Tremelimumab + RT — Patients with an increased CD8+ tumor infiltrating immune cell density and at least clinically stable disease will receive radioimmunotherapy with the PD-L1 Inhibitor Durvalumab and the CTLA4-Inhibitor Tremelimumab (altogether 4 doses q4w including the induction dose) followed by maintenance therapy with Durvalumab (8 additional doses q4w).

SUMMARY:
First-line treatment of locally advanced HNSCC with double checkpoint blockade and radiotherapy dependent on intratumoral CD8+ T cell Infiltration.

DETAILED DESCRIPTION:
This is a single arm, open-label, prospective, non-randomized Phase II clinical trial of locally advanced HNSCC with double checkpoint blockade and radiotherapy dependent on intratumoral CD8+ T cell Infiltration.

All patients will initially be treated with the PD-L1 inhibitor Durvalumab (1500 mg q4w) and the CTLA-4 Inhibitor Tremelimumab (75 mg q4w / since Amendment 3 (01.04.2020): 300 mg absolute dose d5) and one cycle with Cisplatin (30mg/m² d1-3) and Docetaxel (75mg/m² d1). Treatment response will be evaluated clinically by endoscopy with biopsy. Changes of the CD8+ T cell density in the second biopsy compared to the first one before therapy will be used for patient selection. Patients with a stable or decreased CD8+ tumor infiltrating immune cell density or clinical progressive disease will receive standard CRT outside the trial. For these patients toxicity will be monitored until the first dose of the subsequent standard CRT. Patients with an increased CD8+ tumor infiltrating immune cell density and at least clinically stable disease will receive radioimmunotherapy with the PD-L1 Inhibitor Durvalumab and the CTLA4-Inhibitor Tremelimumab (altogether 4 doses q4w including the induction dose) followed by maintenance therapy with Durvalumab (8 additional doses q4w). The primary endpoint is feasibility. Feasibility criteria are receiving the protocol treatment until cycle 6 of antibody treatment and absence of any of the DLT defined in the protocol. A feasibility rate of ≥80% is expected. The efficacy of radioimmunotherapy and predictive character of changes of CD8+ tumor infiltrating immune cells after induction chemo-immunotherapy are further endpoints. The follow up period will be two years after the completion of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization (e.g., HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening Evaluations.
* Age > 18 years at time of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (amend based on specific study)
* Locally advanced HNSCC, UICC stage III-IVB (oral cavity, oropharynx, hypopharynx, supraglottic larynx)
* Histological confirmation of HNSCC (regardless if p16 positive or negative)
* Measureable CD8 density in provided archival tumor tissue
* Body weight >30kg
* Adequate normal organ and marrow function as defined: Haemoglobin ≥ 9.0 g/dL; White blood cells (WBC) ≥ 3,000 per mm3; Platelet count >100,000 per mm3
* Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
* AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal (ULN)
* Creatinine Clearance >40ml/min (calculated from serum creatinine or cystatin C, alternatively 24h urine possible)
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Participation in another clinical study with an investigational product during the last 4 weeks
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Distant metastases
* Prior systemic anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) of the locally advanced HNSCC
* Any other concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment, except the induction chemotherapy in the protocol. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* Prior radiotherapy of HNSCC
* Radiotherapy to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
* Major surgical procedure of the current locally advanced HNSCC (as defined by the Investigator). Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:
* Patients with vitiligo or alopecia areata
* Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients without active disease in the last 5 years may be included but only after consultation with the study physician
* Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for
* Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:
* Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
* Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab + tremelimumab combination therapy.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
* Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period
* Known allergy or hypersensitivity to durvalumab, tremelimumab, cisplatin/carboplatin, docetaxel or any excipient
* Cisplatin/carboplatin induced polyneuropathy or hearing disorder

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Assessment of the number of participants receiving the protocol treatment until cycle 6 of antibody treatment | At the end of cycle 6 of antibody treatment (each cycle is 4 weeks)
  Feasibility means the number of participants receiving the protocol treatment
Assessment of the predictive character of changes of CD8+ tumor infiltrating immune cells after induction chemo-immunotherapy | At Baseline and week 4
  Changes of the CD8+ T cell density in the second biopsy compared to the first one before therapy will be used for patient selection.
Assessment of the absence of any dose-limiting toxicities | At the time of cycle 1 (week 2) to the last cycle 5-12 (up to 2 years)
  Feasibility means the number of dose-limiting toxicities of Grade 3 or higher toxicity that occurs during the trial

SECONDARY OUTCOMES:
Progression free survival | 12 weeks after completion of radiotherapy
  All patients will receive tumor imaging (CT or MRI) 12 weeks after completion of radiotherapy and panendoscopy with biopsy.
Pathologically confirmed response | 12 weeks after completion of radiotherapy
  All patients will receive tumor imaging (CT or MRI) 12 weeks after completion of radiotherapy and panendoscopy with biopsy.
Overall survival | 12 weeks after completion of radiotherapy
  All patients will receive tumor imaging (CT or MRI) 12 weeks after completion of radiotherapy and panendoscopy with biopsy.

OTHER OUTCOMES:
Assessment of predictive value of different tumor infiltrating immune cells and immunological tumor markers. | Baseline (week 0), each cycle is 4 weeks, at the end of cycle 1 (week 2), cycle 2 (week 6), cycle 3 (week 10), cycle 4 (week 14), cycle 5-12 (up to 2 years)
  Longitudinal analysis of the immune phenotype in the peripheral blood.
Assessment of predictive changes of different tumor infiltrating immune cells and immunological tumor markers. | Baseline (week 0), each cycle is 4 weeks, at the end of cycle 1 (week 2), cycle 2 (week 6), cycle 3 (week 10), cycle 4 (week 14), cycle 5-12 (up to 2 years)
  Longitudinal analysis of the immune phenotype in the peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, Prof., Study Chair — Universitätsklinikum Erlangen, Strahlenklinik; Wilfried Budach, Prof., Study Chair — University Düsseldorf; Claus Rödel, Prof., Study Chair — Johann Wolfgang Goethe University Hospital; Markus Hecht, M.D., Principal Investigator — Universitätsklinikum Erlangen; Udo Gaipl, Prof., Study Chair — Universitätsklinikum Erlangen
Locations (7):
- Germany (7):
  - Klinik Chemnitz gGmbH, Chemnitz
  - Dresden, Onkologische Gemeinschaftspraxis, Dresden
  - Düsseldorf, Universitätsklinikum, Klinik für Strahlentherapie und Radiologische Onkologie, Düsseldorf
  - Erlangen, Universitätsklinikum Strahlenklinik, Erlangen
  - Frankfurt, Universitätsklinikum, Klinik für Strahlentherapie und Onkologie, Frankfurt
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beck M, Hartwich J, Eckstein M, Schmidt D, Gostian AO, Muller S, Rutzner S, Gaipl US, von der Grun J, Illmer T, Hautmann MG, Klautke G, Doscher J, Brunner T, Tamaskovics B, Hartmann A, Iro H, Kuwert T, Fietkau R, Hecht M, Semrau S. F18-FDG PET/CT imaging early predicts pathologic complete response to induction chemoimmunotherapy of locally advanced head and neck cancer: preliminary single-center analysis of the checkrad-cd8 trial. Ann Nucl Med. 2022 Jul;36(7):623-633. doi: 10.1007/s12149-022-01744-6. Epub 2022 May 10. PMID 35534690
- [Derived] Hecht M, Eckstein M, Rutzner S, von der Grun J, Illmer T, Klautke G, Laban S, Hautmann MG, Brunner TB, Tamaskovics B, Hinke A, Zhou JG, Frey B, Donaubauer AJ, Becker I, Semrau S, Hartmann A, Balermpas P, Budach W, Gaipl US, Iro H, Gostian AO, Fietkau R. Induction chemoimmunotherapy followed by CD8+ immune cell-based patient selection for chemotherapy-free radioimmunotherapy in locally advanced head and neck cancer. J Immunother Cancer. 2022 Jan;10(1):e003747. doi: 10.1136/jitc-2021-003747. PMID 35078923